CLINICAL TRIAL: NCT00795652
Title: Evidence-based, Distance Treatment for Postpartum Depression, Mom: Managing Our Mood, Part of The Family Help Program
Brief Title: Mom: Managing Our Mood, Part of The Family Help Program
Acronym: MOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3556
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression; Distance therapy; depression; Distance Treatment; Barriers to care
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distance Treatment (Experimental): 50% randomized to receive Distance Treatment for postpartum depression
  Interventions: Behavioral: Distance Treatment for postpartum depression
- Usual Care Services (No Intervention): 50% randomized to receive usual care services for postpartum depression

INTERVENTIONS:
Behavioral: Distance Treatment for postpartum depression — Evidence-based, cognitive behavioural intervention for women with postpartum depression
  Other Names: Family Help Program (listed below: other Modules registered); Pediatric Anxiety (2234a) NCT00267566; Pediatric Disruptive Behaviour (2234b) NCT00267579; Pediatric ADHD NCT00267605; Pediatric Recurrent Headache/abdominal Pain NCT00267618; Pediatric Enuresis NCT00270621; Pediatric Sleep Disorder NCT00338429
  Arms: Distance Treatment

SUMMARY:
The purpose of the MOM: Managing Our Mood Program (part of Family Help) is to evaluate the effectiveness of the Family Help distance intervention compared to usual or standard care typically provided to women with mild to moderate postpartum depression symptomology. This is a single-center trial based at the IWK Health Center. The primary outcome is change in postpartum depression diagnosis.

DETAILED DESCRIPTION:
The Family Help- MOM: Managing Our Mood Program is to deliver, primary care mental health services to mothers in the comfort and privacy of their own home. The purpose of this randomized control trial is to test the effectiveness of the Managing Our Mood (MOM) postpartum depression distance treatment program. This study is a single-centre trial based at the IWK Health Centre, similar to other Family Help Modules.

The goal of this study is to determine the effectiveness of the MOM cognitive-behavioural intervention as an alternative treatment for women suffering from postpartum depression. The intervention is delivered at a distance, using educational materials (handbooks, video-tapes/DVDs, and telephone consultation with a trained paraprofessional coach. Family Help coaches deliver consistent care based on written protocols, with on-going evaluation by a professional team. MOM is not designed to replace specialist care of complex multi-problem mothers.

Eligible participants will be randomly assigned to either active MOM treatment or to the Best Efforts control condition. Those participants assigned to Best Efforts receive printed information about postpartum depression that describes the illness, how it is caused and various treatment options; they are assigned a Coach who books their assessments and is available to answer any questions; they are encouraged to maintain contact and regular care with their family physician or public health nurse for both themselves and their baby. At the end of the 12-month follow-up (one year from randomization), these women will be offered the opportunity to take part in the MOM treatment if they are still depressed.

ELIGIBILITY:
Inclusion Criteria:

* Completed diagnostic measure (SCID), reviewed and signed off by a psychologist
* Participant must meet DSM-IV criteria for postpartum depression
* Significant depressive symptoms that have been present for at least 2 weeks
* Participant must be within 1-12 months postpartum
* Participant must have ready private access to a telephone
* Participant must be between 19-45 years old
* Participant has provided verbal telephone consent
* Participants must speak, read and write in English
* If they are taking medication they must be stabilized (have been on the medication for at least four weeks).

Exclusion Criteria:

* Any condition that in the judgment of the psychologist may interfere with effective delivery of the treatment program (ie, Severe symptomology, challenging diagnostic dilemmas, families who are unmotivated or are in complete chaos)
* Current reports of specific suicidal intentions
* Actively suicidal; suicidal attempts in the previous 6 months
* Participants who are not willing to commit to the demands of treatment
* Participants who have had psychological treatment in the past 6 months for similar problems.
* Participants who have a history of psychotic disorders
* Participants who are cognitively impaired
* Participants who are involved with child protection services
* Participants who have significant substance dependency

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Diagnosis with SCID (Semi-structured diagnostic interview) | baseline, 120, 240, 365

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | baseline, 120, 240, 365
Sheehan Disability Scale | Baseline, 120, 240, 365
Satisfaction measure, designed by the investigator | end of intervention
Beck Depression Inventory-II | baseline, 120, 240 and 365 day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate summary data would be made available but not individual data.

REFERENCES:
- [Background] Lingley-Pottie P, McGrath PJ. Telehealth: a child and family-friendly approach to mental health-care reform. J Telemed Telecare. 2008;14(5):225-6. doi: 10.1258/jtt.2008.008001. PMID 18632994
- [Background] Lingley-Pottie P, McGrath PJ. Distance therapeutic alliance: the participant's experience. ANS Adv Nurs Sci. 2007 Oct-Dec;30(4):353-66. doi: 10.1097/01.ANS.0000300184.94595.25. PMID 18025870
- [Background] Lingely-Pottie P, McGrath PJ. A therapeutic alliance can exist without face-to-face contact. J Telemed Telecare. 2006;12(8):396-9. doi: 10.1258/135763306779378690. PMID 17227604
- [Background] McGrath PJ, Lingley-Pottie P, Emberly DJ, Thurston C, McLean C. Integrated knowledge translation in mental health: family help as an example. J Can Acad Child Adolesc Psychiatry. 2009 Feb;18(1):30-7. PMID 19270846
- [Background] Lingley-Pottie P, McGrath PJ. A paediatric therapeutic alliance occurs with distance intervention. J Telemed Telecare. 2008;14(5):236-40. doi: 10.1258/jtt.2008.080101. PMID 18632997